CLINICAL TRIAL: NCT06563986
Title: Single-arm, Phase II Trial of Trifluridine/Tipiracil (FTD-TPI), Bevacizumab, and Individualized Radioembolization With 166Ho-microspheres in Refractory Metastatic Colorectal Cancer
Brief Title: FTD-TPI, Bevacizumab, and Radioembolization With 166Ho-microspheres in Refractory Metastatic Colorectal Cancer
Acronym: STARLIGHT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Guus Bol, Principal Investigator, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL85987.041.24
Record Dates: First submitted 2024-06-07; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Radioembolization; Trifluridine/Tipiracil; Refractory Metastatic Colorectal Cancer; Radioembolization With 166Ho-microspheres
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention: Systemic treatment (FTD-TPI + bevacizumab) and radioembolization (Experimental): * Individualized dose 166Ho radioembolization, combined with systemic treatment:
  * 35 mg/m2 FTD-TPI on day 1-5 and 8-12 every 4 weeks
  * 5 mg/kg bevacizumab iv. on day 1 and 15 every 4 weeks
  Interventions: Drug: Systemic treatment (FTD-TPI and bevacizumab); Device: Radioembolization with 166-Ho microspheres

INTERVENTIONS:
Drug: Systemic treatment (FTD-TPI and bevacizumab) — Systemic treatment (FTD-TPI and bevacizumab) administration is according to standard clinical practice. Each treatment cycle will be 28 days in duration.
  One treatment cycle consists of the following:
  * Days 1-5: oral intake of FTD-TPI and bevacizumab IV infusion on day 1
  * Days 8-12: oral intake of FTD-TPI
  * Day 15: bevacizumab IV infusion
  Bevacizumab 5.0mg/kg i.v. is repeated every 2 weeks. If toxicity occurs, dose modifications and dose delays should be administered and applied according to standard practice.
Device: Radioembolization with 166-Ho microspheres — Individualized 166Ho radioembolization will be performed via a catheter during angiography. Before the treatment, a scout procedure will be performed to determine individualized 166Ho dose of the treatment. Dosimetry-based treatment planning will be individualized using Q- Suite software.
  In case of bilateral disease, patients will be treated in two procedures to each hemi-liver, separated by 1 month. Before the first procedure, a scout procedure will be performed in which the individualized 166Ho dose of the first and second procedure will be calculated.

SUMMARY:
Extrahepatic disease progression limits clinical efficacy of individualized radioembolization for patients with refractory metastatic colorectal cancer (mCRC). In the same patient population, trifluridine/tipiracil (FTD-TPI) and bevacizumab lead to disease control and overall survival benefit and may be a radiosensitizer.

The purpose of this study is to determine safety, tolerability, and activity of individualized radioembolization with 166Holmium (166Ho)-microspheres combined with FTD-TPI and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable liver dominant mCRC
* Prior therapy with fluoropyrimidine, oxaliplatin, and irinotecan for the treatment of metastatic colorectal cancer and had demonstrated progressive disease or intolerance to their last regimen

  * Patients who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be eligible to enter the study.
  * Patients who refuse oxaliplatin or irinotecan will also be eligible to enter the study.
  * Patients who had received adjuvant chemotherapy and had recurrence during or within 6 months of completion of the adjuvant chemotherapy count the adjuvant therapy as treatment of metastatic colorectal cancer.
* Written informed consent
* Age >=18 years
* Estimated hepatic tumor replacement ≥ 10% and ≤ 50% of total liver volume Eastern Cooperative Oncology Group performance status 0-1
* Adequate organ function as measured by: WBC ≥ 3.0 x 109/L, platelets ≥ 100 x 109/L, absolute neutrophil count > 1.5 x 109/L, Hemoglobin (Hb) > 5 mmol/L (>8.1 g/dL), eGFR ≥ 35 ml/min, Serum transaminases (AST & ALT) ≤ 5 x upper limit of normal (ULN), Total bilirubin ≤ ULN, Albumin > 3 g/dL
* At least one measurable liver lesion according to the PERCIST 1.0

Exclusion Criteria:

* Significant extrahepatic disease, defined as symptomatic extrahepatic disease, more than 10 pulmonary nodules (maximum diameter of each lung metastasis <20mm), and/or peritoneal carcinomatosis.
* Eligible for ablative local treatment of liver metastases (e.g. surgical resection, ablation)
* Lung shunt >20 Gy, as calculated using scout dose SPECT/CT
* Absorbed tumor dose <90 Gy when dosing at a maximum average absorbed normal liver dose
* Other malignancy confounding prognosis
* Receipt of chemotherapy within 28 days prior to study treatment
* Previous or current treatment with radioembolization
* Major surgery within 28 days or incompletely healed surgical incision before starting study therapy
* Any serious comorbidity preventing the safe administration of anti-VEGF antibody treatment. This includes uncontrolled hypertension or treatment with ≥3 antihypertensive drugs, arterial (cerebro)vascular event within the past 6 months, history of severe bleeding, history of GI perforation, or presence of fistulae
* Any serious and/or chronic liver disease preventing the safe administration of radio- embolization
* Uncorrectable extrahepatic deposition of scout dose activity; activity in the falciform ligament, portal lymph nodes and gallbladder is accepted
* Pregnancy or breastfeeding
* Body weight over 150 kg (because of maximum table load)
* Known severe allergy for intravenous contrast fluids
* Participation to another investigational study which may compromise any endpoint of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Hepatic objective response rate (hORR) (PERCIST 1.0) | Evaluated every 8 weeks after the start of treatment until 1 year after the start of treatment or until disease progression, whichever comes first.
  Hepatic objective response rate (hORR) will be assessed by Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) 1.0.

SECONDARY OUTCOMES:
Hepatic objective response rate (hORR) (RECIST 1.1) | Evaluated every 8 weeks after the start of treatment until 1 year after the start of treatment or until disease progression, whichever comes first.
  Hepatic objective response rate (hORR) will be assessed by Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
Overall and extra-hepatic ORR (RECIST 1.1) | Evaluated every 8 weeks after the start of treatment until 1 year after the start of treatment or until disease progression, whichever comes first.
  Overall and extra-hepatic ORR will be assessed by RECIST 1.1.
Overall and extra-hepatic ORR (PERCIST 1.0) | Evaluated every 8 weeks after the start of treatment until 1 year after the start of treatment or until disease progression, whichever comes first.
  Overall and extra-hepatic ORR will be assessed by PERCIST 1.0.
Serious adverse events (SAE's) | Evaluated every 8 weeks after start treatment during the first half year. The collection period will start from the first day of the first treatment cycle until 180 days thereafter.
  The occurrence of any (suspected unexpected) serious adverse event (SAE) that is possibly, probably or definitely related to the combined treatment.
Grade ≥3 adverse events (CTCAE 5.0) | Evaluated every 8 weeks after start treatment during the first half year. The collection period will start from the first day of the first treatment cycle until 180 days thereafter.
  The rate of grade ≥3 adverse events (CTCAE 5.0).
Occurrence of radioembolization-induced liver disease (REILD) | Evaluated every 8 weeks after start treatment during the first half year.
  Radioembolization-induced liver disease (REILD) is defined as a total bilirubin increase to grade ≥3 or higher according to the CTCAE v5.0, in combination with ascites and low albumin, developing at least 2 weeks after radioembolization and up to 4 months after radioembolization, in the absence of tumor progression or biliary obstruction.
Radioembolization related vascular events | Evaluated every 8 weeks after start treatment during the first half year.
  Number of participants with a vascular event (dissection, pseudo-aneurism, thrombus etc.) that is possibly, probably or definitely related to the radioembolization.
Dose reductions, dose delays of FTD-TPI | Evaluated during the first two cycles (each cycle is 28 days).
  The frequency of dose reductions and dose delays of FTD-TPI during the first 2 cycles.
Radioembolization completion rate | Evaluated immediately after the radioembolization treatment.
  Defined as the successful treatment of both hemi-livers (in case of bilateral disease) according to the individualized treatment plan designed at the scout dose.
Progression free survival (PFS) | Evaluated every 8 weeks after the start of treatment until 1 year after the start of treatment or until disease progression, whichever comes first.
  PFS is defined as time from the first day of the first treatment cycle to progression of disease or death, whichever occurs first. Progression of disease is based on tumor response as observed on radiographic imaging according to RECIST 1.1.
Overall survival (OS) | Evaluated once per year until the end of the study (the end of study is defined as six months after the first day of the first treatment cycle (each cycle is 28 days) of the 36th evaluable participant).
  OS is defined as the time from the first day of the first treatment cycle to the date of death. Patients still alive at the analysis cut-off date are censored at the last date known to be alive. OS will be collected for all patients from the Personal Records Database (BRP), yearly during the duration of the study.

OTHER OUTCOMES:
Dosimetry scout + post treatment 1 and 2 | Evaluated immediately after the radioembolization treatment.
  To evaluate biodistribution / dosimetry using CT and quantitative SPECT both for scout dose imaging and post-treatment imaging. Tumor dose and normal liver dose will be calculated for each hemi-liver in the scout procedure and two post treatment scans.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No